CLINICAL TRIAL: NCT01499810
Title: Study of Efficacy and Safety of Radiofrequency Sympathetic Renal Denervation for Treatment of Drug Resistant Hypertension
Brief Title: Efficacy and Safety of Radiofrequency Renal Denervation in Drug Resistant Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Stanislav Pekarskiy, Principal Investigator, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Hypertension
Keywords: Hypertension; Radiofrequency Catheter Ablation; Renal Artery; Sympathetic Nerve Block
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal denervation (Experimental): All eligible patients undergo bilateral radiofrequency sympathetic renal denervation using endocardial ablation system: after standard renal angiography using femoral access a small size endocardial ablation catheter (5-6 F, 4 mm electrode) is inserted into renal artery and 4-8 point ablations are performed consecutively from distal part to aorta with 3-4 mm step and 90 degrees rotation on the upper, lower, front and back aspects of the artery to get circumferential coverage, then the procedure is repeated on the other side.
  Interventions: Procedure: Bilateral radiofrequency sympathetic renal denervation

INTERVENTIONS:
Procedure: Bilateral radiofrequency sympathetic renal denervation — Bilateral radiofrequency sympathetic renal denervation is performed as percutaneous transluminal radiofrequency (RF) ablation of neural pathways in the renal artery walls and surrounding tissue using standard equipment for RF ablation of cardiac electrical pathways
  Other Names: Transcatheter renal denervation; Percutaneous radiofrequency ablation of renal nerves

SUMMARY:
Single-center, single group study of the efficacy and safety of transcatheter renal denervation for treatment of patients with essential hypertension uncontrolled despite combined pharmacotherapy including 3 or more hypotensive drugs one of which is a diuretic. Bilateral transcatheter renal denervation will be performed on the top of existed pharmacotherapy. Change in blood pressure (BP), left ventricle (LV) mass, carotid artery thickness, renal artery blood flow and renal function, will be assessed at 6 and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 80 years at time of randomization
* Informed consent
* Treatment with full doses of 3 or more anti-hypertensive medications of different classes, of which one is a diuretic.
* Office Systolic BP (SBP) ≥ 160 mmHg or Diastolic BP (DBP) ≥ 100 mmHg

Exclusion Criteria:

* An estimated glomerular filtration rate (eGFR) of < 30 mL/min/1.73 m2
* Ambulatory Blood Pressure Monitoring (ABPM) 24 hour average SBP < 135 mmHg or DBP < 85 mmHg
* Symptomatic(secondary) hypertension
* Severe renal artery stenosis or renal arteries abnormalities
* Individual is pregnant, nursing or planning to be pregnant
* Severe hepatic dysfunction
* Any other clinically important renal, hematological, metabolic, neurological, gastrointestinal, hepatic or pulmonary disorders or dysfunctions preventing study participation (investigator's assessment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislav E Pekarskiy, MD, Principal Investigator — Institute of Cardiology, Siberian Branch of the Russian Academy of Medical Sciences
Locations (1):
- Institute of Cardiology, Siberian Branch of Russian Academy of Medical Sciences, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] S. Pekarskiy, A. Baev, V. Mordovin, T. Ripp, G. Semke, V. Lichikaki, E. Sitkova, A. Krylov, S. Popov, R. Karpov, Renal denervation by endocardial ablation system, European Heart Journal, Volume 34, Issue suppl_1, 1 August 2013, 3788, https://doi.org/10.1093/eurheartj/eht309.3788
- [Derived] Ripp TM, Mordovin VF, Pekarskiy SE, Ryabova TR, Zlobina MV, Baev AE, Anfinogenova Y, Popov SV. Predictors of Renal Denervation Efficacy in the Treatment of Resistant Hypertension. Curr Hypertens Rep. 2015 Dec;17(12):90. doi: 10.1007/s11906-015-0603-8. PMID 26482895

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive patients admitted to our clinic for resistant hypertension were evaluated for eligibility according to selection criteria pre-defined in protocol of this study
Pre-assignment Details: 83 patients with true resistant hypertension were identified, 12 rejected the intervention, 11 were excluded for anatomical reasons: atherosclerosis of renal arteries - 7, multiple narrow renal arteries - 2, fibromuscular dysplasia (FMD) - 1 and aneurysm of renal artery - 1. Finally 53 subjects were included and undergone renal denervation
Groups:
- Renal Denervation: All eligible patients undergone bilateral radiofrequency sympathetic renal denervation using endocardial ablation system: after standard renal angiography using femoral access a small size endocardial ablation catheter (5-6 F, 4 mm electrode) was inserted into renal artery and 4-10 point ablations were performed consecutively from distal part to aorta with 3-4 mm step and 90 degrees rotation on the upper, lower, front and back aspects of the artery to get circumferential coverage, then the procedure is repeated on the other side.
  Bilateral radiofrequency sympathetic renal denervation: Bilateral radiofrequency sympathetic renal denervation was performed as percutaneous transluminal radiofrequency (RF) ablation of neural pathways in the renal artery walls and surrounding tissue using standard equipment for RF ablation of cardiac electrical pathways
Period: Overall Study
Arm/Group | Renal Denervation
Started | 53
Completed | 41
Not Completed | 12
Not completed — Lost to Follow-up | 10
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Renal Denervation
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 52
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in Office Systolic BP
Time Frame: from baseline to 12 months
Population: All patients who completed 12 month assessment according to the protocol.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 41
mmHg | -31.1 (24.0)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

2. Primary Outcome: Number of Serious Adverse Events
Description: A number of first occurrences (within the study period) of any of the following: death, end-stage renal disease, an embolic event resulting in end-organ damage, major bleeding event, renal artery thrombosis, new renal artery stenosis, other serious cardiovascular complications if their relation to the study treatment is assessed at least as possible.
Time Frame: from baseline to 12 months
Measure: Number; unit: Events
Arm/Group | Renal Denervation
Number analyzed (Participants) | 41
Events | 0

3. Secondary Outcome: Change in Office Diastolic BP
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 41
mmHg | -15.4 (15.6)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

4. Secondary Outcome: Change in Mean 24-h Systolic BP
Time Frame: from baseline to 12 months
Population: Number of participants assessed at 12 months minus 1 participant with unsatisfactory ambulatory blood pressure monitoring (ABPM) record
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -11.9 (15.9)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

5. Secondary Outcome: Change in Mean 24-h Diastolic BP
Time Frame: from baseline to 12 months
Population: Number of participants assessed at 12 months minus 1 participant with unsatisfactory ABPM record
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -7.6 (10.1)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

6. Secondary Outcome: Change in Office Systolic BP
Time Frame: from baseline to 6 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 46
mmHg | -27.1 (24.8)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

7. Secondary Outcome: Change in Office Diastolic BP
Time Frame: from baseline to 6 month
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 46
mmHg | -13.3 (15.7)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

8. Secondary Outcome: Change in Mean 24-h Systolic BP
Time Frame: from baseline to 6 months
Population: Number of participants assessed at 6 months minus 2 participants with unsatisfactory ABPM records
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | -10.3 (15.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

9. Secondary Outcome: Change in Mean 24-h Diastolic BP
Time Frame: from baseline to 6 months
Population: Number of participants assessed at 6 months minus 2 participants with unsatisfactory ABPM record
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | -6.2 (9.0)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

10. Secondary Outcome: Change in Echocardiographic Left Ventricular Mass
Time Frame: from baseline to 6 months
Population: Number of participants assessed by echocardiography (EchoCG ) at 6 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Renal Denervation
Number analyzed (Participants) | 45
g | -10.1 (71.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.35, t-test, 2 sided — threshold for statistical significance p<0.05

11. Secondary Outcome: Change in Echocardiographic Left Ventricular Mass
Time Frame: from baseline to 12 months
Population: Number of participants assessed by EchoCG at 12 months
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
g | -14.6 (61.4)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.12, t-test, 2 sided — threshold for statistical significance p<0.05

12. Secondary Outcome: Change in Mean Daytime Systolic BP
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 45
mmHg | -11.0 (16.5)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.00007, t-test, 2 sided — threshold for statistical significance p<0.05

13. Secondary Outcome: Change in Mean Daytime Diastolic BP
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 45
mmHg | -6.7 (10.2)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.00009, t-test, 2 sided — threshold for statistical significance p<0.05

14. Secondary Outcome: Change in Mean Daytime Systolic BP
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -12.3 (16.7)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.00004, t-test, 2 sided — threshold for statistical significance p<0.05

15. Secondary Outcome: Change in Mean Daytime Diastolic BP
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -7.7 (11.4)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — threshold for statistical significance p<0.05

16. Secondary Outcome: Change in Mean Nighttime Systolic BP
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | -9.2 (16.7)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.0007, t-test, 2 sided — threshold for statistical significance p<0.05

17. Secondary Outcome: Change in Mean Nighttime Diastolic BP
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | -5.0 (9.5)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — threshold for statistical significance p<0.05

18. Secondary Outcome: Change in Mean Nighttime Systolic BP
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -11.2 (18.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided — threshold for statistical significance p<0.05

19. Secondary Outcome: Change in Mean Nighttime Diastolic BP
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -7.3 (11.1)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided — threshold for statistical significance p<0.05

20. Secondary Outcome: Change in Mean Nighttime Systolic BP Dipping
Description: Mean nighttime BP dipping is a relative difference: absolute difference between mean daytime and mean nighttime BP values divided by mean daytime BP value
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: percentages
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
percentages | -0.4 (8.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.57, t-test, 2 sided — threshold for statistical significance p<0.05

21. Secondary Outcome: Change in Mean Nighttime Diastolic BP Dipping
Description: as for outcome 20
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: percentages
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
percentages | -1.1 (9.0)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.54, t-test, 2 sided — threshold for statistical significance p<0.05

22. Secondary Outcome: Change in Mean Nighttime Systolic BP Dipping
Description: as for outcome 20
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: difference between percentages
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
difference between percentages | -0.23 (8.73)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.87, t-test, 2 sided — threshold for statistical significance p<0.05

23. Secondary Outcome: Change in Mean Nighttime Diastolic BP Dipping
Description: as for outcome 20
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: percentages
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
percentages | 0.47 (10.23)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.77, t-test, 2 sided — threshold for statistical significance p<0.05

24. Secondary Outcome: Change in Daytime Systolic BP Variability
Description: daytime/nighttime BP variability is a standard deviation of BP values measured respectively during daytime/nighttime periods in course of ambulatory BP monitoring (ABPM)
Time Frame: from baseline to 12 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -1.4 (4.5)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.06, t-test, 2 sided — threshold for statistical significance p<0.05

25. Secondary Outcome: Change in Daytime Diastolic BP Variability
Description: daytime/nighttime BP variability is a standard deviation of BP values measured respectively during daytime/nighttime periods in course of ambulatory BP monitoring
Time Frame: from baseline to 12 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -1.0 (3.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.07, t-test, 2 sided — threshold for statistical significance p<0.05

26. Secondary Outcome: Change in Nighttime Systolic BP Variability
Description: as for outcome 25
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -0.83 (5.27)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.32, t-test, 2 sided — threshold for statistical significance p<0.05

27. Secondary Outcome: Change in Nighttime Diastolic BP Variability
Description: as for outcome 25
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 40
mmHg | -1.03 (4.13)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.12, t-test, 2 sided — threshold for statistical significance p<0.05

28. Secondary Outcome: Change in Daytime Systolic BP Variability
Description: as for outcome 25
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | -0.2 (4.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.72, t-test, 2 sided — threshold for statistical significance p<0.05

29. Secondary Outcome: Change in Daytime Diastolic BP Variability
Description: as for outcome 25
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | 0.4 (3.0)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.37, t-test, 2 sided — threshold for statistical significance p<0.05

30. Secondary Outcome: Change in Nighttime Systolic BP Variability
Description: as for outcome 25
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | -0.01 (5.0)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.99, t-test, 2 sided — threshold for statistical significance p<0.05

31. Secondary Outcome: Change in Nighttime Diastolic BP Variability
Description: as for outcome 25
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
mmHg | 0.2 (4.8)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.76, t-test, 2 sided — threshold for statistical significance p<0.05

32. Secondary Outcome: Change in Serum Creatinine
Time Frame: from baseline to 1 week
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Renal Denervation
Number analyzed (Participants) | 51
micromol/l | 2.4 (9.8)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.08, t-test, 2 sided — threshold for statistical significance p<0.05

33. Secondary Outcome: Change in Serum Creatinine
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Renal Denervation
Number analyzed (Participants) | 45
micromol/l | -1.6 (11.3)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.35, t-test, 2 sided — threshold for statistical significance p<0.05

34. Secondary Outcome: Change in Serum Creatinine
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: micromol/l
Arm/Group | Renal Denervation
Number analyzed (Participants) | 41
micromol/l | 1.9 (13.9)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.22, t-test, 2 sided — threshold for statistical significance p<0.05

35. Secondary Outcome: Change in Casual Proteinuria
Description: Change of protein concentration in morning urine sample
Time Frame: from baseline to 1 week
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Renal Denervation
Number analyzed (Participants) | 39
g/l | -0.04 (0.2)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.29, t-test, 2 sided — threshold for statistical significance p<0.05

36. Secondary Outcome: Change in Casual Proteinuria
Description: Change of protein concentration in morning urine sample
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
g/l | -0.005 (0.2)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.89, t-test, 2 sided — threshold for statistical significance p<0.05

37. Secondary Outcome: Change in Casual Proteinuria
Description: Change of protein concentration in morning urine sample
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Renal Denervation
Number analyzed (Participants) | 39
g/l | 0.05 (0.09)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.65, t-test, 2 sided — threshold for statistical significance p<0.05

38. Secondary Outcome: Change in Specific Gravity of Urine
Description: Change of specific gravity of morning urine sample
Time Frame: from baseline to 1 week
Measure: Mean (Standard Deviation); unit: no specific units
Arm/Group | Renal Denervation
Number analyzed (Participants) | 39
no specific units | -0.38 (7.9)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.76, t-test, 2 sided — threshold for statistical significance p<0.05

39. Secondary Outcome: Change in Specific Gravity of Urine
Description: Change of specific gravity of morning urine sample
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: no specific units
Arm/Group | Renal Denervation
Number analyzed (Participants) | 44
no specific units | 1.0 (7.1)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.35, t-test, 2 sided — Repeated measures analysis

40. Secondary Outcome: Change in Specific Gravity of Urine
Description: Change of specific gravity of morning urine sample
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: no specific units
Arm/Group | Renal Denervation
Number analyzed (Participants) | 41
no specific units | -0.07 (5.7)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.92, t-test, 2 sided — threshold for statistical significance p<0.05

41. Secondary Outcome: Change in Renal Resistive Index Measured by Doppler Flowmetry in Left Main Renal Artery
Description: Resistive index calculated as relative difference between assessed by ultrasound Doppler maximal and minimal blood flow velocities, i.e. absolute difference between maximal and minimal blood flow velocities divided by maximal flow velocity
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: difference between two ratios
Arm/Group | Renal Denervation
Number analyzed (Participants) | 45
difference between two ratios | -0.008 (0.055)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.32, t-test, 2 sided — threshold for statistical significance p<0.05

42. Secondary Outcome: Change in Renal Resistive Index Measured by Doppler Flowmetry in Right Main Renal Artery
Description: as for outcome 41
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: difference between two ratios
Arm/Group | Renal Denervation
Number analyzed (Participants) | 45
difference between two ratios | 0.010 (0.075)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.40, t-test, 2 sided — threshold for statistical significance p<0.05

43. Secondary Outcome: Change in Resistive Index Measured by Renal Doppler Flowmetry in Left Main Renal Artery
Description: as for outcome 41
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: difference between ratios
Arm/Group | Renal Denervation
Number analyzed (Participants) | 37
difference between ratios | -0.011 (0.06)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.17, t-test, 2 sided — threshold for statistical significance p<0.05

44. Secondary Outcome: Change in Resistive Index Measured by Renal Doppler Flowmetry in Right Main Renal Artery
Description: as for outcome 41
Time Frame: from baseline to 12 months
Measure: Mean (Standard Deviation); unit: difference between ratios
Arm/Group | Renal Denervation
Number analyzed (Participants) | 37
difference between ratios | -0.019 (0.07)
Statistical Analysis 1: Comparison: Renal Denervation; Repeated measures analysis; Test type: Superiority or Other; p = 0.014, t-test, 2 sided — threshold for statistical significance p<0.05

45. Secondary Outcome: Change in Ultrasound Intima Media Thickness of Carotid Artery
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

46. Secondary Outcome: Change in Ultrasound Intima Media Thickness of Carotid Artery
Time Frame: from baseline to 12 months
Reporting Status: Not Posted

47. Secondary Outcome: Change in Arterial Stiffness
Description: Change of cardio-ankle vascular index(CAVI) assessed by vascular screening device VaSera VS1000 (name of the model)
Time Frame: from baseline to 12 months
Reporting Status: Not Posted

48. Secondary Outcome: Change in Arterial Stiffness
Description: Change of cardio-ankle vascular index(CAVI) assessed by vascular screening device VaSera VS1000
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

49. Secondary Outcome: Change in Morning Surge of BP
Time Frame: from baseline to 12 months
Reporting Status: Not Posted

50. Secondary Outcome: Change in Morning Surge of BP
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Renal Denervation
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 3/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=53)
Pospunctional pseudoaneurysm of femoral artery (Injury, poisoning and procedural complications) | 3 (3) — Small hematoma communicating with the lumen of femoral artery occurred as a result of percutaneous punction of the femoral artery in course the procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No